CLINICAL TRIAL: NCT03036943
Title: An Open-labelled Study to Characterise Fluciclovine (18F) Uptake Measured by positRon emissiON Tomography In Breast cancER
Brief Title: Fluciclovine (18F) Imaging of Breast Cancer
Acronym: FRONTIER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OCTO_078
Record Dates: First submitted 2016-12-09; First posted 2017-01-31 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fluciclovine (18F) PET/CT (Experimental)
  Interventions: Radiation: Fluciclovine

INTERVENTIONS:
Radiation: Fluciclovine — Fluciclovine (18F) PET/CT scan completed >= 48 hours prior to surgical resection for breast cancer
  Other Names: 18F; FACBC

SUMMARY:
The purpose of this study is to find out what a new amino acid-based PET agent, fluciclovine (18F), can tell us about breast cancer biology (how it grows and develops), and quantify the differences in fluciclovine (18F) uptake between breast cancer subtypes. This will inform further work to investigate its use in breast cancer management.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven breast cancer (invasive ductal or ductal carcinoma in situ (DCIS)) measuring ≥ 1.5cm

   * Tumour size should be based on the longest diameter measured on ultrasound, mammogram or MRI performed within 2 months prior to enrolment.
2. No prior treatment for breast cancer.
3. Female, Age >= 40 years.
4. The patient is willing and able to comply with the protocol scheduled visits and examinations for the duration of the study. Women of childbearing potential must follow contraception guidance given as standard of care at breast cancer diagnosis.
5. Written (signed and dated) informed consent.

Exclusion Criteria:

1. Pregnant or breastfeeding women
2. Major surgery or significant traumatic injury within four weeks prior to enrolment.
3. Treatment with any other investigational agent, or participation in another interventional clinical study within 4 weeks prior to enrolment.
4. Multifocal breast cancer (defined as more than two tumours, either unilateral or bilateral).
5. Known hypersensitivity to fluciclovine (18F) or any of its constituents.
6. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor study candidate or could interfere with protocol compliance or the interpretation of study results.
7. Any other active malignancy or any previous diagnosis of melanoma.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Tumour standardised uptake values (SUV) in invasive breast cancer, classified by molecular type, on fluciclovine (18F) PET imaging. | From PET/CT scan commencing approx 30 seconds after fluciclovine (18F) administration

SECONDARY OUTCOMES:
Amino acid transporter (AAT) and related growth pathway expression levels quantitatively assessed by immunohistochemistry using the H-score method, and correlated to fluciclovine (18F) uptake (SUV). | From tumour samples taken during standard of care surgery 48 hours or greater after PET/CT scan
Tumour metabolite levels characterized by fold change compared to metabolite levels in the adjacent normal tissue, and correlated to fluciclovine (18F) uptake. | From tumour samples taken during standard of care surgery 48 hours or greater after PET/CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Harris, Prof, Principal Investigator — University of Oxford
Locations (1):
- Churchill Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scott NP, Teoh EJ, Flight H, Jones BE, Niederer J, Mustata L, MacLean GM, Roy PG, Remoundos DD, Snell C, Liu C, Gleeson FV, Harris AL, Lord SR, McGowan DR. Characterising 18F-fluciclovine uptake in breast cancer through the use of dynamic PET/CT imaging. Br J Cancer. 2022 Mar;126(4):598-605. doi: 10.1038/s41416-021-01623-3. Epub 2021 Nov 18. PMID 34795409